CLINICAL TRIAL: NCT06271954
Title: The Relationship Between Emotion Regulation and Psychiatric Disorder in Youth - From a Psychosocial Developmental Aspect.
Brief Title: The Relationship Between Emotion Regulation and Psychiatric Disorder in Youth
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, Tzu-Yu Liu, occpatioal therapist, Chang Gung Memorial Hospital
Other Study IDs: 202300096A3
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Major Depressive Disorder; Anxiety Disorder; Attention Deficit Hyperactivity Disorder (ADHD); Adjustment Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders; Attention Deficit Disorder with Hyperactivity; Adjustment Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- control: (1) Understanding the content of the questionnaire. (2) Healthy adolescents aged 15 to less than 18 years and healthy adults aged 18 to 24 years.
- experimental: (1) Understanding the content of the questionnaire. (2) Adolescents aged 15 to less than 18 years and adults aged 18 to 24 years. (3) Diagnosed with major depressive disorder, anxiety disorder, attention deficit hyperactivity disorder (ADHD), or adjustment disorder according to DSM-5.

SUMMARY:
According to the increasing worldwide prevalence rate of psychiatric disorders in youth, the mental health of youth is becoming more and more important.

Taiwan's Ministry of Health and Welfare reported the clibing suicide rate of youth in past five years and showed the prevention work and related intervention for youth's mental health was noteable. The definition of emotion regulation was "consists of the extrinsic and intrinsic processes responsible for monitoring, evaluating, and modifying emotional reactions, especially their intensive and temporal features, to accomplish one's goals." Emotion regulation strategies including "rumination", "avoidance", "suppression", "Problem-solving", "reappraisal", "acceptance", "social support", and "distraction".

Previous studies had examined the relationship between emotion regulation and mental health in youth; maladaptive emotion regulation would increase the individual's depressive and anxiety symptoms. Carstensen proposed social emotion theory in 1995 Selectivity theory (SST) refers to the need for emotion regulation, which activates Social participation in late adulthood. SST assumes that young people are more interested in social interaction behaviors related to information seeking and building self-concept. characteristics of youth affected by many normative challenges such as adolescence, school transitions, and more complex social Landscape; Adaptive emotion regulation will reduce risk of clinical emotion attacks of illness, especially depression and anxiety.To explore the relationship between emotion regulation and mental health from a psychosocial developmental aspect, we focused on the interaction between individual and environment. Compared with the previous generation, most youths of this generation were participating in social activities and building up interpersonal relationships through the internet, suggesting the internet was an important social context.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for the control group are as follows: (1) Understanding the content of the questionnaire. (2) Healthy adolescents aged 15 to less than 18 years and healthy adults aged 18 to 24 years.

The inclusion criteria for the experimental group are:

1. Understanding the content of the questionnaire.
2. Adolescents aged 15 to less than 18 years and adults aged 18 to 24 years.
3. Diagnosed with major depressive disorder, anxiety disorder, attention deficit hyperactivity disorder (ADHD), or adjustment disorder according to DSM-5.

Exclusion Criteria:

* The exclusion criteria for the experimental group are diagnoses of:

  1. organic brain injury
  2. schizophrenia
  3. autism spectrum disorder according to DSM-5.

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Use the Cognitive Emotion Regulation Questionnaire (CERQ) to assess subjective emotion regulation patterns in community healthy young people's emotion regulation experiences and expressions, and measure personal emotion regulation patterns related to mental health.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2025-03-26 (Estimated); Study Completion 2025-03-26 (Estimated)

PRIMARY OUTCOMES:
The Difference and Similarity in Emotional Regulation Strategy Patterns between Western and Eastern Countries. | Each respondent interviews and fills out questionnaires, which takes about 20minutes.
  To examine the cultural difference in emotion regulation strategies, we applied CERQ(Cognitive Emotion Regulation Questionnaire) to measure the cognitive regulation pattern of the Taiwanese and compared it with research articles that reported the CERQ results in six European countries and China.
  Cognitive Emotion Regulation Questionnaire (CERQ). The CERQ includes nine positive/negative adaptive emotion regulation strategies: self-blame, rumination, Blaming others, catastrophizing, acceptance, positive refocusing, refocus on planning, positive reappraisal, putting into perspective ), each strategy subscale contains 4 questions, a total of 36 questions, and is answered in the form of a five-point scale. Subjects describe each question and circle the options that are consistent with their own situation (never, rarely, sometimes , often, always), each item ranges from 1 "never" to 5 "always", one point per question, no reverse questions.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang-Geng Medical Foundation Chang-Geng Memorial Hospital, Keelung, Taiwan